CLINICAL TRIAL: NCT04267393
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multiple-Dose Phase 2 Study to Evaluate the Efficacy and Safety of BMS-986263 in Adults With Compensated Cirrhosis From Nonalcoholic Steatohepatitis (NASH)
Brief Title: Safety and Effectiveness of BMS-986263 in Adults With Compensated Cirrhosis (Liver Disease) From Nonalcoholic Steatohepatitis (NASH)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial terminated because of lack of efficacy in the short term acute phase.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM025-017; 2019-003932-22 (EudraCT Number); U1111-1241-4762 (Other: UTN Number)
Record Dates: First submitted 2020-02-11; First posted 2020-02-12 (Actual); Results first posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Nonalcoholic Steatohepatitis (NASH)
Keywords: Nonalcoholic Steatohepatitis; Liver Disease; NASH; Compensated cirrhosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose A BMS-986263 (Experimental)
  Interventions: Drug: BMS-986263
- Dose B BMS-986263 (Experimental)
  Interventions: Drug: BMS-986263
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BMS-986263 — Specified dose on specified days
  Arms: Dose A BMS-986263; Dose B BMS-986263
Other: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this randomized study is to assess safety and effectiveness of BMS-986263 in adults with compensated cirrhosis (chronic liver disease) from nonalcoholic steatohepatitis (fatty liver disease) (NASH).

ELIGIBILITY:
Inclusion Criteria:

* Participants with liver biopsy fibrosis score stage 4 (NASH CRN) performed within 12 months
* Men and women must agree to follow methods of contraception

Exclusion Criteria:

* Worsening liver disease or any disease might compromise participant safety in the opinion of the investigator
* Known immunocompromised status or any disease or condition which might compromise participant safety
* Prior exposure to BMS-986263
* Clinically relevant abnormal physical examination, vital signs, ECG, or clinical laboratory tests
* Hepatic decompensation

Other protocol-defined inclusion/exclusion criteria apply

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2024-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (111):
- United States (29):
  - Arizona Clinical Trials - Tucson, Chandler, Arizona
  - Local Institution - 0173, Chandler, Arizona
  - The Institute for Liver Health-The Institute for Liver Health, Chandler, Arizona
  - Local Institution, Phoenix, Arizona
  - Local Institution - 0140, La Jolla, California
  - Local Institution - 0205, Lancaster, California
  - GastroIntestinal BioSciences, Los Angeles, California
  - Local Institution - 0143, Redwood City, California
  - Florida Research Institute, Lakewood Rch, Florida
  - Local Institution - 0024, Leesburg, Florida
  - Local Institution - 0061, Miami, Florida
  - Local Institution - 0025, Winter Park, Florida
  - Local Institution - 0121, Iowa City, Iowa
  - Local Institution - 0150, Baltimore, Maryland
  - Local Institution, Fall River, Massachusetts
  - Local Institution - 0077, Kansas City, Missouri
  - Local Institution - 0186, Omaha, Nebraska
  - Research Foundation of SUNY - University of Buffalo, Buffalo, New York
  - NYU Langone Health-Department of Medicine, New York, New York
  - Local Institution, New York, New York
  - Local Institution - 0206, Morehead City, North Carolina
  - Local Institution - 0177, Philadelphia, Pennsylvania
  - Local Institution - 0017, Philadelphia, Pennsylvania
  - University Diabetes & Endocrine Consultants, Chattanooga, Tennessee
  - Local Institution - 0171, Dallas, Texas
  - Local Institution - 0109, Houston, Texas
  - Local Institution, McAllen, Texas
  - Local Institution - 0013, San Antonio, Texas
  - Local Institution - 0122, Richmond, Virginia
- Argentina (4):
  - Local Institution - 0089, Ciudad de Buenos Aires, Buenos Aires
  - Local Institution - 0126, San Juan Bautista, Buenos Aires
  - Local Institution - 0209, Quilmes, Buenos Aires F.D.
  - Local Institution - 0059, Buenos Aires
- Belgium (3):
  - Local Institution - 0009, Edegem
  - Local Institution - 0006, Ghent
  - Local Institution - 0133, Leuven
- Brazil (9):
  - Local Institution - 0083, Salvador, Estado de Bahia
  - Local Institution - 0182, Bento Gonçalves, Rio Grande do Sul
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0187, Barretos, São Paulo
  - Local Institution - 0188, Botucatu, São Paulo
  - Local Institution, Ribeirão Preto, São Paulo
  - Local Institution - 0196, São Bernardo do Campo, São Paulo
  - Local Institution - 0120, São Paulo
  - Local Institution, São Paulo
- Canada (2):
  - Local Institution - 0128, Victoria, British Columbia
  - Local Institution - 0097, Toronto, Ontario
- France (7):
  - Local Institution - 0094, Lyon
  - Local Institution - 0031, Nice
  - Local Institution - 0101, Paris
  - Local Institution - 0105, Paris
  - Local Institution - 0137, Strasbourg
  - Local Institution - 0029, Vandœuvre-lès-Nancy
  - Local Institution - 0202, Créteil, Île-de-France Region
- Germany (9):
  - Local Institution - 0082, Frankfurt am Main, Hesse
  - Local Institution - 0091, Berlin
  - Local Institution - 0099, Essen
  - Local Institution - 0096, Hanover
  - Local Institution - 0073, Kiel
  - Local Institution - 0194, Lübeck
  - Local Institution - 0071, Mainz
  - Local Institution - 0060, Munich
  - Local Institution - 0204, Trier
- Israel (4):
  - Local Institution - 0056, Haifa
  - Local Institution - 0076, Petah Tikva
  - Local Institution - 0058, Ramat Gan
  - Local Institution - 0057, Tel Aviv
- Italy (5):
  - Local Institution - 0054, Bologna
  - Azienda Ospedaliera Universitaria Di Messina G. Martino-D.A.I. Medicina Interna, Messina
  - Local Institution - 0115, Palermo
  - Local Institution - 0051, Pisa
  - Local Institution, Rome
- Japan (16):
  - Local Institution - 0200, Tōon, Ehime
  - Local Institution - 0048, Kurume, Fukuoka
  - Local Institution - 0049, Sapporo, Hokkaido
  - Local Institution - 0127, Shiwagun Yahabatyo, Iwate
  - Local Institution - 0075, Yokohama, Kanagawa
  - Local Institution - 0155, Matsumoto, Nagano
  - Local Institution - 0111, Kashihara, Nara
  - Local Institution - 0163, Sakai, Osaka
  - Local Institution - 0125, Bunkyō, Tokyo
  - Local Institution - 0138, Minato-ku, Tokyo
  - Local Institution - 0199, Aomori
  - Local Institution - 0193, Gifu
  - Local Institution - 0026, Hiroshima
  - Local Institution - 0135, Kagoshima
  - Local Institution - 0131, Kyoto
  - Local Institution - 0132, Yamagata
- Local Institution - 0012, San Juan, Puerto Rico
- South Korea (3):
  - Local Institution - 0093, Incheon, Incheon-gwangyeoksi [Incheon]
  - Local Institution - 0066, Seodaemun-gu
  - Local Institution - 0090, Seoul
- Spain (9):
  - Local Institution - 0040, Barcelona
  - Local Institution - 0080, Madrid
  - Local Institution - 0039, Madrid
  - Local Institution - 0038, Madrid
  - Local Institution - 0036, Málaga
  - Local Institution - 0037, Santander
  - Local Institution - 0041, Seville
  - Local Institution - 0035, Valencia
  - Local Institution - 0043, Valencia
- Switzerland (2):
  - Local Institution - 0102, Lugano, Canton Ticino
  - Local Institution - 0074, Bern
- Taiwan (3):
  - Local Institution - 0001, Kaohsiung City
  - Local Institution, Taipei
  - Local Institution - 0004, Taoyuan District
- United Kingdom (5):
  - Local Institution - 0011, Nottingham, Nottinghamshire
  - Local Institution - 0034, Hull
  - Local Institution - 0124, Liverpool
  - Local Institution - 0005, London
  - Local Institution, Southampton

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo
- Treatment 1: BMS-986263 45mg QW
- Treatment 2: BMS-986263 90mg QW
Period: Randomization
Arm/Group | Placebo | Treatment 1 | Treatment 2
Started | 40 | 42 | 42
Completed (= Randomized and Treated) | 39 | 41 | 42
Not Completed | 1 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Administrative Reasons by Sponsor | 0 | 1 | 0
Period: Treatment Period
Arm/Group | Placebo | Treatment 1 | Treatment 2
Started | 39 | 41 | 42
Completed | 36 | 35 | 35
Not Completed | 3 | 6 | 7
Not completed — Adverse Event | 0 | 2 | 3
Not completed — Participant Withdrew Consent | 0 | 0 | 1
Not completed — Administrative Reasons by Sponsor | 3 | 4 | 3

BASELINE CHARACTERISTICS:
Population: All Randomized Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Total
Number analyzed (Participants) | 40 | 42 | 42 | 124
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.9 (8.56) | 58.9 (6.76) | 60.0 (8.65) | 59.3 (7.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 25 | 25 | 72
  Male | 18 | 17 | 17 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 13 | 18 | 53
  Not Hispanic or Latino | 7 | 18 | 17 | 42
  Unknown or Not Reported | 11 | 11 | 7 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 11 | 9 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 34 | 31 | 32 | 97
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve ≥ 1 Stage Improvement in Liver Fibrosis (NASH CRN Fibrosis Score), as Determined by Liver Biopsy After 12 Weeks of Treatment.
Description: Percentage of participants who achieve ≥ 1 stage improvement in liver fibrosis (NASH CRN Fibrosis Score), as determined by liver biopsy after 12 weeks of treatment.
  For the NASH CRN Fibrosis Score, fibrosis is staged on a 0 to 4 scale: 0 (none); 1 (perisinusoidal or periportal fibrosis); 2 (perisinusoidal and portal/periportal fibrosis); 3 (bridging fibrosis); 4 (cirrhosis).
  Responder is defined as achieved >=1 stage improvement in liver fibrosis (NASH CRN Fibrosis Score) as determined by liver biopsy from baseline to week 12/early treatment termination (ETT).
Time Frame: 12 Weeks
Population: Modified Intent to Treat Population (mITT)
Measure: Number; unit: Percentage
Arm/Group | Placebo | Treatment 1 | Treatment 2
Number analyzed (Participants) | 39 | 41 | 42
Percentage | 20.5 | 12.2 | 7.1

2. Secondary Outcome: Percentage of Participants Who Achieve ≥ 1 Stage Improvement in Liver Fibrosis (NASH CRN Fibrosis Score) With no Worsening of NASH After 12 Weeks of Treatment.
Description: Percentage of participants who achieve ≥ 1 stage improvement in liver fibrosis (NASH CRN Fibrosis Score) with no worsening of NASH after 12 weeks of treatment.
  For the NASH CRN Fibrosis Score, fibrosis is staged on a 0 to 4 scale: 0 (none); 1 (perisinusoidal or periportal fibrosis); 2 (perisinusoidal and portal/periportal fibrosis); 3 (bridging fibrosis); 4 (cirrhosis).
Time Frame: 12 Weeks
Population: mITT population
Measure: Number; unit: Percentage
Arm/Group | Placebo | Treatment 1 | Treatment 2
Number analyzed (Participants) | 39 | 41 | 42
Percentage | 20.5 | 12.2 | 4.8

3. Secondary Outcome: Percentage of Participants Who Achieve ≥ 2 Stage Improvement in Liver Fibrosis (NASH CRN Fibrosis Score) With no Worsening of NASH After 12 Weeks of Treatment.
Description: Percentage of participants who achieve ≥ 2 stage improvement in liver fibrosis (NASH CRN Fibrosis Score) with no worsening of NASH after 12 weeks of treatment.
  For the NASH CRN Fibrosis Score, fibrosis is staged on a 0 to 4 scale: 0 (none); 1 (perisinusoidal or periportal fibrosis); 2 (perisinusoidal and portal/periportal fibrosis); 3 (bridging fibrosis); 4 (cirrhosis).
Time Frame: 12 Weeks
Population: mITT Population
Measure: Number; unit: Percentage
Arm/Group | Placebo | Treatment 1 | Treatment 2
Number analyzed (Participants) | 39 | 41 | 42
Percentage | 2.6 | 0 | 0

4. Secondary Outcome: Percentage of Participants Who Achieve ≥ 1 Stage Improvement in Liver Fibrosis (Modified Ishak Score) After 12 Weeks of Treatment.
Description: Percentage of participants who achieve ≥ 1 stage improvement in liver fibrosis (modified Ishak score) after 12 weeks of treatment.
  A modified Ishak scoring system (0 to 6 scale) was originally developed to grade portal-based liver fibrosis associated with viral hepatitis. The modified Ishak system has been adapted to grade central-based liver fibrosis associated with NASH, and it also uses a 0 to 6 scale:
  0: No fibrosis
  1. perisinusoidal or periportal fibrosis
  2. perisinusoidal and portal/periportal fibrosis
  3. bridging fibrosis with linkage of < 50% of vascular structures (portal and centrilobular)
  4. bridging fibrosis with linkage of > 50% of vascular structures (portal and centrilobular)
  5. early or incomplete cirrhosis
  6. established or advanced cirrhosis
Time Frame: 12 Weeks
Population: mITT Population
Measure: Number; unit: Percentage
Arm/Group | Placebo | Treatment 1 | Treatment 2
Number analyzed (Participants) | 39 | 41 | 42
Percentage | 30.8 | 26.8 | 21.4

5. Secondary Outcome: Percentage of Participants Who Achieve ≥ 2 Stage Improvement in Liver Fibrosis (Modified Ishak Score) After 12 Weeks of Treatment.
Description: Percentage of participants who achieve ≥ 2 stage improvement in liver fibrosis (modified Ishak score) after 12 weeks of treatment.
  A modified Ishak scoring system (0 to 6 scale) was originally developed to grade portal-based liver fibrosis associated with viral hepatitis. The modified Ishak system has been adapted to grade central-based liver fibrosis associated with NASH, and it also uses a 0 to 6 scale:
  0: No fibrosis
  1. perisinusoidal or periportal fibrosis
  2. perisinusoidal and portal/periportal fibrosis
  3. bridging fibrosis with linkage of < 50% of vascular structures (portal and centrilobular)
  4. bridging fibrosis with linkage of > 50% of vascular structures (portal and centrilobular)
  5. early or incomplete cirrhosis
  6. established or advanced cirrhosis
Time Frame: 12 Weeks
Population: mITT Population
Measure: Number; unit: Percentage
Arm/Group | Placebo | Treatment 1 | Treatment 2
Number analyzed (Participants) | 39 | 41 | 42
Percentage | 10.3 | 4.9 | 4.8

6. Secondary Outcome: Mean Change From Baseline in CPA After 12 Weeks of Treatment
Description: Change from baseline in CPA after 12 weeks of treatment.
  Assessment of collagen proportionate area(CPA) is a method by which the amount (percentage) of collagen in stained tissue sections is analyzed using morphometric image analysis. This allows for a quantitative assessment of fibrosis. Percentage of fat in stained tissue sections is also analyzed using morphometric image analysis.
Time Frame: 12 Weeks
Population: Total number of evaluable participants are those who have both baseline and Week 12/ETT biopsy available
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Placebo | Treatment 1 | Treatment 2
Number analyzed (Participants) | 35 | 32 | 27
Percentage | -3.67 (1.861) | -0.35 (1.374) | -3.67 (1.973)

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) and Treatment Emergent Serious Adverse Events (TESAE)
Description: An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does have a causal relationship with this treatment.
Time Frame: From First Treatment to end of Follow up (36 weeks)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2
Number analyzed (Participants) | 39 | 41 | 42
Participants
  TEAE | 24 | 33 | 34
  TESAE | 1 | 1 | 2

8. Secondary Outcome: Number of Participants With Clinically Significant Changes in Clinical Laboratory Values.
Description: Investigators must document their review of each laboratory safety report. A central laboratory will perform the analyses and will provide reference ranges for these tests.
  clinical laboratory assessments analyzed: Hematology, Blood Chemistry, Urinalysis and a Metabolic Panel.
Time Frame: From First Treatment to end of Follow up (36 weeks)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2
Number analyzed (Participants) | 39 | 41 | 42
Participants | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vitals Signs.
Description: Includes body temperature, respiratory rate, blood pressure, and heart rate. Blood pressure and heart rate should be measured after the participant has been resting quietly for at least 5 minutes.
Time Frame: From First Treatment to end of Follow up (36 weeks)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2
Number analyzed (Participants) | 39 | 41 | 42
Participants | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Changes in Physical Examination Findings.
Description: Physical examination includes body weight, height, and BMI (height and BMI calculation at screening only).
Time Frame: From First Treatment to end of Follow up (36 weeks)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2
Number analyzed (Participants) | 39 | 41 | 42
Participants | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram Readings.
Description: Number of Participants with clinically significant changes in electrocardiogram readings.
Time Frame: From First Treatment to end of Follow up (36 weeks)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2
Number analyzed (Participants) | 39 | 41 | 42
Participants | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Clinically Significant Changes in BMD.
Description: Bone Mineral Density(BMD) will be measured by a dual-energy X-ray absorptiometry (DXA) Scan.
Time Frame: From First Treatment to end of Follow up (36 weeks)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2
Number analyzed (Participants) | 39 | 41 | 42
Participants | 0 | 0 | 0

13. Secondary Outcome: Plasma Concentration of BMS-986263 Components at the End of 12 Weeks or ETT.
Description: Plasma concentrations of BMS-986263 components: siRNA, DPD, HEDC, and S104.
Time Frame: 12 Weeks
Population: All participants who receive at least 1 dose of BMS-986263 and have any available concentration-time data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Placebo | Treatment 1 | Treatment 2
Number analyzed (Participants) | 0 | 42 | 42
ng/mL
  siRNA: number analyzed (Participants) | 0 | 17 | 19
  siRNA |  | 38.9 (151) | 72.9 (169)
  DPD: number analyzed (Participants) | 0 | 28 | 42
  DPD |  | 519 (45.2) | 1138 (80.7)
  HEDC: number analyzed (Participants) | 0 | 28 | 28
  HEDC |  | 25.1 (51.8) | 59.0 (58.8)
  S104: number analyzed (Participants) | 0 | 3 | 6
  S104 |  | 4.16 (141) | 3.68 (50.7)

ADVERSE EVENTS:
Time Frame: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication Adverse Events and Serious Adverse Events: (From first dose to last dose + 24 week follow up): Approximately 36 Weeks All-Cause mortality (From randomization to end of study): Approximately 42 Weeks.
Groups:
- Placebo: Placebo QW
Arm/Group | Placebo | Treatment 1 | Treatment 2
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/41 | 0/42
Serious Adverse Events (participants affected / at risk) | 1/39 | 1/41 | 2/42
Other Adverse Events (participants affected / at risk) | 17/39 | 24/41 | 29/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=39) | Treatment 1 (N=41) | Treatment 2 (N=42)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Infected cyst (Infections and infestations) | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=39) | Treatment 1 (N=41) | Treatment 2 (N=42)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 2 | 1
Asthenia (General disorders) | 2 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 4
COVID-19 (Infections and infestations) | 4 | 4 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 17 | 22
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0
Headache (Nervous system disorders) | 4 | 4 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT04267393/Prot_SAP_000.pdf